CLINICAL TRIAL: NCT02876939
Title: Proprioception and Sensorimotor Control in Hereditary Sensory and Autonomic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-00530
Record Dates: First submitted 2016-08-05; First posted 2016-08-24 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Atunomic Neuropathy
Keywords: Hereditary Sensory Neuropathy; Autonomic Neuropathy; Familial Dysautonomia; proprioception; motor control; sensory nervous system.; HSAN III; IKBKAP gene mutation
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies; Dysautonomia, Familial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HSAN III (Experimental)
  Interventions: Other: kinesiology tape around the hip, knee and ankle joints; Other: No kinesiology tape around the hip, knee and ankle joints
- Control Subjects (Active Comparator)
  Interventions: Other: kinesiology tape around the hip, knee and ankle joints; Other: No kinesiology tape around the hip, knee and ankle joints

INTERVENTIONS:
Other: kinesiology tape around the hip, knee and ankle joints — We will also demonstrate that taping the skin increases the central representation of cutaneous afferent input in HSAN III.
Other: No kinesiology tape around the hip, knee and ankle joints — Investigators will demonstrate that taping the skin increases the central representation of cutaneous afferent input in HSAN III.

SUMMARY:
This project comprises three sets of physiological studies - testing eight specific hypotheses - that will contribute new knowledge on proprioception and motor control in a genetic disorder that affects specific components of the sensory nervous system.

I: To investigate the neurophysiological basis for disturbed motor control in Hereditary sensory and autonomic neuropathy (HSAN) III II: To investigate the effects of enhancing cutaneous feedback on motor control in HSAN III III: To investigate the cortical representation of proprioceptive inputs in HSAN III

DETAILED DESCRIPTION:
HSAN III patients (n=15) and healthy control subjects (n=15) will lay supine on an MRI bed and a tungsten microelectrode inserted percutaneously into a muscle or cutaneous fascicle of the right common peroneal nerve at the fibular head, according to standard techniques employed by Prof Macefield. Neural activity will be acquired, RMS-processed (200 ms) and analysed on computer. The subject's head will be tightly enclosed in a standard clinical 32-channel SENSE head coil and headphones will be provided to minimize noise and to allow communication with the subject. The subject will be placed in the bore of a 3T whole-body scanner for 60-90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed genetic diagnosis of HSAN III will be recruited from the Dysautonomia Center at NYU

Exclusion Criteria:

* homeless
* active drug or alcohol dependence
* evidence of neurological disorder or diabetes
* exposure to neurotoxic drugs that in the investigator's opinion may compromise results
* Pregnant women

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Measurement of gait in HSAN III | 120 Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Horacio Kaufmann, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States